CLINICAL TRIAL: NCT06218888
Title: A Phase II Clinical Study of the Efficacy and Safety of Tislelizumab Combined With Fruquintinib and Chidamide in the Treatment of Unresectable or Advanced Microsatellite Stabilized (MSS/pMMR) Colorectal Cancer With Liver Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TFC
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — tislelizumab; HMPL-013; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with fruquintinib and Chidamide (Experimental): The treatment option for the chidamide + tislelizumab +fruquibtinib is 200 mg of tislelizumab IV Drip Q3W, 30 mg of chidamide PO BIW, and fruquibtinib 3mg PO Q3W until loss of clinical benefit or development of intolerable toxicity
  Interventions: Drug: Tislelizumab; Drug: Fruquintinib; Drug: Chidamide

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg，D1, Q3W
Drug: Fruquintinib — Fruquintinib 3mg ,D1-D14, Q3W
Drug: Chidamide — Chidamide 30mg

SUMMARY:
To explore the Efficacy and Safety of Tislelizumab combined with fruquintinib and Chidamide in the treatment of unresectable or advanced microsatellite stabilized (MSS/pMMR) colorectal cancer with liver metastases

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ≤ 75 years old.
* Expected survival time ≥ 18 weeks.
* Diagnosis of pMMR confirmed by PCR for microsatellite stability (MSS) or low microsatellite instability (MSI-L), or by immunohistochemistry for DNA mismatch repair (MMR) proteins, including MLH1, MSH2, MSH6 and PMS2 protein expression, which result in no protein deletion.
* Subjects with histologically and/or cytologically confirmed locally advanced unresectable or metastatic colorectal adenocarcinoma with liver metastasis (excluding adenosquamous carcinoma mixed with other pathological types).
* ECOG PS score is in the range of 0~1.
* Failure of previous treatment with fluorouracil, oxaliplatin, and irinotecan based chemotherapy, with imaging evidence (such as CT scans) or clinical evidence (such as cytological reports of new ascites or pleural effusion) demonstrating disease progression during or after treatment, or discontinuation of treatment due to toxicity intolerance.
* Subjects having adequate organ and bone marrow functions with laboratory test values within 7 days prior to enrollment meeting the following requirements, as follows:

  1. Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥ 100×109/L; hemoglobin level (HGB) ≥ 9.0 g/dL.
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN in subjects without liver metastases, and ALT and AST ≤ 5.0 × ULN in subjects with liver metastases; serum albumin ≥ 25 g/L.
  3. Renal function: serum creatinine (Cr) ≤ 1.5 x ULN. 4) Patients with routine urine results showing urine protein <2+ or routine urine testing showing urine protein ≥ 2+ at baseline should undergo 24-hour urine collection and 24-hour urine protein quantification < 1 g.

  5) Coagulation function: international normalized ratio (INR) ≤ 1.5×ULN and activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

Exclusion Criteria:

* Prior exposure to any anti-PD-1 antibody, anti-PD-L1 antibody, HDAC inhibitor, or irinotecan.
* Receiving any investigational drug within 4 weeks prior to the first dose of the study drug.
* Concurrent participation in another interventional clinical study, except in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study.
* Receiving the last dose of antitumor therapy (chemotherapy, targeted therapy, tumor immunotherapy, or tumor embolization) within 3 weeks prior to the first dose.
* Receiving radiotherapy within 4 weeks prior to the first dose.
* Patients who have received radiotherapy more than 4 weeks prior to the first dose with any radiotherapy-related toxic reactions, such as radiation pneumonia, radiation hepatitis, radiation enteritis, including clinical symptoms only, or requiring glucocorticoid therapy.
* Use of immunosuppressive drugs within 4 weeks prior to the first dose, excluding topical glucocorticoids by nasal spray, inhalation or other routes or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/day prednisone or equivalent doses of other glucocorticoids).
* Receiving live attenuated vaccine within 4 weeks prior to the first dose or planning to receive during the study period.
* Major surgical procedure (craniotomy, thoracotomy or open heart surgery) or unhealed wound, ulcer or fracture within 4 weeks prior to the first dose.
* Presence of toxicity (excluding alopecia, non-clinically significant and asymptomatic laboratory abnormalities) from prior antineoplastic therapy not recovered to ≤ grade 1 by NCI common terminology criteriafor adverse events (CTCAE) Version 5.0 (NCI CTCAE Version 5.0) prior to the first dose.
* Known presence of symptomatic CNS metastases and/or carcinomatous meningitis. Subjects with prior treatment for brain metastases may participate in the study provided that the brain metastases have remained stable for at least 4 weeks prior to the first dose of study treatment; and that neurological symptoms have recovered to ≤ grade 1 by NCI CTCAE version 5.0.
* Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are allowed. A known history of primary immunodeficiency. For patients with only positive autoimmune antibodies, the presence of autoimmune diseases should be confirmed at the discretion of the investigator.
* Patients who are known to have active tuberculosis and are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to the first dose.
* Known to have interstitial lung disease requiring steroid hormone therapy.
* Known to have acute or chronic active hepatitis B (HBsAg positive and HBV DNA ≥ 200 IU/mL or ≥ 103 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive).
* Infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive), known to be infected with syphilis.
* Severe infections that are in the active phase or poorly controlled in clinical practice. Serious infection, including but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia, within 4 weeks prior to the first dose.
* Significant malnutrition, such as the need for intravenous supplemental nutrient solutions; except for malnutrition corrected more than 4 weeks prior to the first dose.
* Symptomatic congestive heart failure (New York Heart Association class II-IV); symptomatic or poorly controlled arrhythmias.
* Uncontrolled arterial hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) even with standard treatment.
* Any arterial thromboembolic event including myocardial infarction, pulmonary embolism, and unstable angina within 6 months prior to enrollment.
* A history of deep vein thrombosis or any other serious thromboembolism (implantable IV port or catheter-derived thrombosis, or superficial vein thrombosis is not considered "serious" thromboembolism) within 3 months prior to enrollment.
* Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or more severe cirrhosis.
* A history of gastrointestinal perforation and/or fistula in the previous 6 months; a history of peptic ulcer, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, abdominal abscess, or long-term chronic diarrhea. Post-intestinal stent implantation.

  -> 3 loose stools per day at baseline, suggesting a predisposition to colon or small bowel disease with uncontrollable symptoms.
* A history of allergy or known intolerance to atropine sulfate or loperamide or the appropriate antiemetic in combination with FOLFIRI.
* Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary reactions to cancer and can lead to higher medical risk and/or uncertainty in survival evaluation.
* A known history of inherited bleeding tendency disorders or coagulation disorders.
* Any life-threatening bleeding event within the previous 3 months, including the need for blood transfusion therapy, surgical or local treatment, or ongoing drug therapy.
* A high risk of bleeding as determined by the investigators: cirrhosis with severe esophagogastric fundic varices, intermittent or persistent non-fatal bleeding events (including but not limited to intermittent bloody stools or positive occult blood due to primary intestinal lesions, intermittent hemoptysis due to pulmonary metastases).

Cerebrovascular accident (including transient ischemic attack) in the previous 6 months.

* Use of aspirin (>325 mg/day) or other NSAIDs known to inhibit platelet function for 10 consecutive days within 10 days prior to the first dose.
* Treatment with oral or parenteral anticoagulants or thrombolytics for 10 consecutive days within 10 days prior to the first dose. However, prophylactic use of anticoagulants is allowed.
* Pleural fluid, ascites, and pericardial effusion with clinical symptoms or requiring drainage, except for small amounts of pleural fluid, small amounts of ascites, and small amounts of pericardial effusion without clinical symptoms on imaging only.
* A history of other primary malignancies, except: malignancies in complete response for at least 2 years prior to enrollment and requiring no other treatment during the study period; adequately treated non-melanoma skin cancer or malignant freckled nevus with no evidence of disease recurrence; adequately treated carcinoma in situ with no evidence of disease recurrence.
* A known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Known to be allergic to any monoclonal antibody component.
* Female subjects in the pregnancy or lactating period.
* A history of alcohol or drug abuse.
* Other acute or chronic illnesses, psychiatric disorders, or abnormal laboratory test values that may result in the following outcomes: increasing the risk associated with study participation or study drug administration, or interfering with the interpretation of study results and, at the investigator's discretion, classifying the patient as ineligible for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | Around 2 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Around 2 years
  Time from enrollment to disease progression or death from any cause
Disease Control Rate (DCR) | Around 2 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR), partial response (PR) or stable disease (SD) according to RECIST 1.1.